CLINICAL TRIAL: NCT00903565
Title: A Prospective Study for the Assessment of Recurrence Risk in Stage II Colon Cancer Patients Using ColoPrint
Acronym: PARSC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-060-CR
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Colon Cancer
Keywords: genomic profiling; gene expression; ColoPrint; adenocarcinoma colon; recurrence risk assessment; prospective
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to enroll 785 eligible stage II colon cancer patients in order to validate the performance of ColoPrint in estimating 3-year relapse rate.

Secondary objectives include comparing the objective risk assessment results from the prognostic profile (ColoPrint) to both the risk assessment based on the ASCO criteria, as well as the Investigator's independent assessment. As this is the first prospective study of ColoPrint, this study will also address the logistics and quality assurance of using ColoPrint in clinical practice.

Patient treatment is at the discretion of the physician, adhering to National Comprehensive Cancer Network (NCCN)-approved regimens or a recognized alternative.

The enrollment period will be 6 years. It is expected that 1800 to 2400 patients will be enrolled in order to obtain 785 analysable stage II samples from eligible patients. Approximately 25-35 clinical sites will be involved worldwide.

The statistical analysis will be performed by Agendia and an independent research institute or hospital.

Study Design Extension Study:

This will be a prospective study to measure the impact of ColoPrint on adjuvant treatment in stage 2 colorectal cancer patients. After surgery the tumor sample will be shipped in RNA Retain to Agendia. The online Clinical Report Form (CRF) 0 will be completed to document if the patient fulfils the inclusion criteria. Baseline clinical data and the patient and physician chemotherapy intention, patient's perceived recurrence risk and decisional conflict without knowing the ColoPrint result will be entered in CRF 1. After completion of CRF1 the ColoPrint result is released. CRF2 will be completed after the final treatment decision has been made.

This CRF will capture the patient and physician chemotherapy intention, patient's perceived recurrence risk and decisional conflict, impact of ColoPrint and the actual treatment the patient will receive. CRF3 will be completed 12 months after enrolment and will capture the patient status, patient's perceived recurrence risk and decisional conflict. CRF4 and 5 will be completed 3 and 5 years after surgery and will capture the patient status. A sample size of 210 stage 2 colon cancer patients is required to detect a 10% overall treatment change (5% significance and 90% power).

Reporting of the Results:

Blinded Study; The ColoPrint results will not be reported to the physician and/or patient at the time of enrolment. All samples will be stored in a freezer until 550-575 eligible stage II patients have been enrolled. Samples will then be analyzed in one batch in a blinded fashion from the clinical results.

Extension Study; The ColoPrint results will be reported to the physician and patient after CRF1 has been completed.

DETAILED DESCRIPTION:
Primary Objective • To validate the performance of ColoPrint in estimating the 3-year relapse rate in patients with stage II colorectal cancer.

Secondary Objectives

• To assess the feasibility of using the ColoPrint test in the clinical setting.

* To compare the risk assessment in stage II patients using the ColoPrint profile vs a clinical risk assessment based on 1) Investigator's assessment of risk and 2) ASCO high-risk recommendations (T4 lesions, perforation / obstruction, inadequate node sampling (less than 12 nodes) or poorly differentiated histology).
* To establish the proportion of low-risk and high-risk ColoPrint profiles in stage II colorectal cancer patients in various countries.
* To investigate therapy as a potential confounding factor for ColoPrint results.
* To assess the performance of ColoPrint in estimating the 3-year relapse rate in patients with stage III colorectal cancer.
* To compare the performance of ColoPrint vs the clinical risk assessment in estimating the 5-year relapse rate.
* Assess the impact of ColoPrint on adjuvant chemotherapy treatment decisions in stage 2 colorectal cancer patients
* Compare the ColoPrint results from fresh RNARetain colorectal tumor specimens to the matched formalin-fixed paraffin-embedded tissue (FFPE) colon tumor specimens for concordance.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* adenocarcinoma of the colon or rectum
* stage II-III, planned to be treated with radical surgery

Exclusion Criteria:

* prior malignancy with the exception of basal cell carcinoma or cervical dysplasia
* any neo-adjuvant therapy
* synchronous tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from participating hospitals worldwide
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2008-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To validate the performance of ColoPrint in estimating the 3-year relapse rate in patients with stage II colorectal cancer. | The enrolment period will be 6 years

SECONDARY OUTCOMES:
• To assess the feasibility of using the ColoPrint test in the clinical setting. | The enrolment period will be 6 years
• To compare the risk assessment in stage II patients using the ColoPrint profile vs a clinical risk assessment | The enrolment period will be 6 years
• To establish the proportion of low-risk and high-risk ColoPrint profiles in stage II colorectal cancer patients in various countries. | The enrolment period will be 6 years
• To investigate therapy as a potential confounding factor for ColoPrint results. | The enrolment period will be 6 years
• To assess the performance of ColoPrint in estimating the 3-year relapse rate in patients with stage III colorectal cancer. | The enrolment period will be 6 years
• To compare the performance of ColoPrint vs the clinical risk assessment in estimating the 5-year relapse rate. | The enrolment period will be 6 years
• Assess the impact of ColoPrint on adjuvant chemotherapy treatment decisions in stage 2 colorectal cancer patients | The enrolment period will be 6 years
• Compare the ColoPrint results from fresh RNARetain colorectal tumor specimens to the matched formalin-fixed paraffin-embedded tissue (FFPE) colon tumor specimens for concordance. | The enrolment period will be 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Salazar, MD, Principal Investigator — Institut Català D´Oncologia, L'Hospitalet Barcelona; John L Marshall, MD, Principal Investigator — Chief, Division of Hematology/Oncology, Georgetown University Hospital Washington
Locations (35):
- United States (17):
  - Glendale Memorial Hospital, Glendale, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Sutter Roseville Medical Center /Research, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - UC Davis Cancer Center, Sacramento, California
  - Scripps Cancer Center, San Diego, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Atlanta Colon and Rectal Surgery, Riverdale, Georgia
  - Albert Einstein College of Medicine, Montefiore Medical Center, The Bronx, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Franciscan Research Center, Tacoma, Washington
- Austria (3):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Krankenhaus der Elisabethinen, Linz
  - Medical University of Vienna, Vienna
- University of Hong Kong/ Queen Mary Hospital, Hong Kong, China
- Odense Universitetshospital, Odense, Denmark
- CRLC Val d'Aurelle-Paul Lamarque, Montpellier, France
- Klinikum Rechts Der Isar, Munich, Germany
- Matsuda Hospital, Hamamatsu, Japan
- Netherlands (4):
  - Medisch Centrum Alkmaar, Alkmaar
  - Medisch Spectrum Twente, Enschede
  - Westfriesgasthuis, Hoorn
  - LUMC, Leiden
- Spain (2):
  - Vall d' Hebron University Hospital, Barcelona
  - IDIBELL Institut Catala d'Oncologia (ICO), L'Hospitalet de Llobregat
- Immunology Akademiska sjukhuset/ University Hospital, Uppsala, Sweden
- Kantonsspital Baden, Baden, Switzerland
- United Kingdom (2):
  - Norfolk and Norwich University Hospital, Norwich
  - University of Oxford, Oxford

REFERENCES:
- See also: Related Info — http://www.agendia.com